CLINICAL TRIAL: NCT06365970
Title: Phase II Study of Niraparib and Dostarlimab for Patients With MMR-D/MSI-H Colorectal Cancers: A Proof of Concept Study
Brief Title: Niraparib and Dostarlimab for Patients With MMR-D/MSI-H Colorectal Cancers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Per drug sponsor request.
Sponsor: Ibrahim Halil Sahin (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Ibrahim Halil Sahin, Assistant Professor of Medical oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 23-056
Record Dates: First submitted 2024-03-29; First posted 2024-04-15 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: MMR-D/MSI-H Colorectal Cancers
Keywords: PARP inhibitor; MRE11 deficiency; Immune checkpoint inhibitor; Homologous recombination defect; HRD; MSI-H/MMR-D Colorectal cancer; Niraparib; Dostarlimab
MeSH Terms: interventions — niraparib; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib + Dostarlimab (Experimental): Niraparib: 300/200 mg daily (weight-based dosing*)
  Dostarlimab: 500 mg Q3 weeks
  *Weight-based dosing: Patients weighing ≥77 kg (≥170 lbs) AND a platelet count ≥150,000/mcL, the niraparib dose is determined to be 300 mg taken orally once daily continuously in combination with dostarlimab 500 mg every 3 weeks.
  Patients weighing <77 kg (<170 lbs) OR with a platelet count <150,000/mcL, the niraparib dosage will be 200 mg taken orally, once daily continuously in combination with dostarlimab 500 mg every 3 weeks (Q3W)
  Interventions: Drug: Niraparib; Drug: Dostarlimab

INTERVENTIONS:
Drug: Niraparib — An anti-cancer medication that helps to repair DNA when it becomes damaged, known as a PARP inhibitor.
  Other Names: Zejula
Drug: Dostarlimab — An anti-cancer medication that is a programmed death receptor-1 -blocking monoclonal antibody.
  Other Names: Jemperli

SUMMARY:
The second line of therapy for patients with MSI-H CRC who experience disease progression on anti-PD1 based therapies is not well defined and there is an unmet need for research for patients with anti-PD1 refractory MSI-H CRC. This study will examine the combination of niraparib and dostarlimab for a synergistic antitumor effect for patients with MSI-H CRC.

DETAILED DESCRIPTION:
In this single-arm phase II study, the clinical effectiveness of niraparib in combination with dostarlimab will be investigated for patients with MSI-H colorectal cancer who had disease progression on anti-PD1-based therapy. This study aims to leverage MRE11 deficiency and other HR pathway alterations by using Niraparib and also aims to create potential synergetic effect between dostarlimab with niraparib combination to induce clinically meaningful antitumor benefit. Patients with advanced stage MSI-H CRC who progressed on first line anti-PD1 +/- anti-CTLA4 based therapy will be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed mismatch repair deficient or microsatellite instability high advanced stage colorectal cancer
2. Measurable disease per RECIST v1.1
3. ECOG 0 to 2
4. Age ≥ 18 years
5. Able to swallow oral medication (tablets).
6. Progression on prior anti-PD1 ± anti-CTLA4 therapy.
7. Adequate organ function based on the following lab assessments:

   1. ANC must be ≥ 1500/mm3.
   2. Platelet count must be ≥ 100,000/mm3.
   3. WBC count ≥ 2.5 × 109 /L
   4. Hemoglobin must be ≥ 9 g/dL.
   5. Alkaline phosphatase ≤ 2.5× upper limit of normal (ULN) with the exception of patients with documented liver or bone metastases who should have ALP ≤ 5.0× ULN.
   6. AST and ALT≤ 2.5× ULN with the exception of patients with documented liver metastases who may have AST and/or ALT ≤ 5.0× ULN.
   7. International normalized ratio (INR) ≤ 1.5 x ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless receiving treatment with therapeutic anticoagulation.
   8. Total bilirubin ≤ 1.5× ULN (≤3× ULN if Gilbert syndrome present)
   9. Serum albumin ≥ 2.8 g/dL or 28 g/L
   10. Creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault equation.
8. Patient who experienced progression of disease on prior anti-PD1 ± Anti-CTLA in the adjuvant and neoadjuvant settings are eligible to be enrolled in this trial without requirement of a second line of immunotherapy for advanced stage disease.
9. Women of childbearing potentials must use a contraceptive method that is highly effective (with a failure rate of <1% per year), from the screening visit through at least 120 days after the last dose of study treatment and agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period.
10. Men must agree to use adequate contraception for the duration of trial participation and for 4 months after the last dose of study drugs. Men must also agree to not donate sperm. Men must agree to use adequate contraception for the duration of trial participation and for 4 months after the last dose of study drugs. Men must also agree to not donate sperm.

Exclusion Criteria:

1. More than 2 lines of systemic therapy (excluding adjuvant therapy)
2. Prior oxaliplatin based chemotherapy for metastatic disease. This excludes adjuvant oxaliplatin. Patients who received oxaliplatin based chemotherapy for metastatic disease before determination of MMR-D/MSI-H status (due to test turn-around time) can be enrolled if they received 4 or less cycle of oxaliplatin treatment (each cycle is one dose).
3. More than 1 line of anti-PD1 based therapy.
4. History of severe hypersensitivity to anti-PD1 monoclonal antibodies
5. Prior PARPi
6. Progression on platinum-based chemotherapy
7. Active autoimmune disease requiring immune suppression except following conditions:

   1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone without an active complication are eligible for the study.
   2. Patients with well controlled Type 1 diabetes mellitus who are actively on an insulin regimen are eligible for the study.
   3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      * Disease is well controlled at baseline and requires only topical corticosteroids. - No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
8. Active untreated brain metastasis (patients treated brain metastasis within 4 weeks can be enrolled)
9. Any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.
10. Received colony-stimulating factors (e.g., granulocyte macrophage colony-stimulating factor or recombinant erythropoietin) within 4 weeks.
11. Previously or are currently participating in a treatment study of an investigational agent within 4 weeks of the first dose of therapy preceding the study.
12. Received live vaccine within 30 days of planned start of study randomization. Study patients can be vaccinated against Corona virus disease 2019 (COVID-19) using vaccines authorized via the appropriate regulatory mechanisms. Note: messenger ribonucleic acid (mRNA) and adenoviral-based COVID-19 vaccines are considered nonlive. If COVID-19 vaccine is administered at any time, the date, name of the COVID-19 vaccine anatomic location, must be entered in the eCRF.
13. Hypersensitivity to the components of niraparib or the formulation excipients.
14. Undergone major surgery within 4 weeks of starting the first dose of study treatment or have not recovered from any effects of any major surgery.
15. Have a second primary malignancy. Exceptions are the following:

    1. Adequately treated nonmelanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast, Stage I Grade 1 endometrial carcinoma
    2. Other solid tumors and lymphomas (without bone marrow involvement) diagnosed ≥5 years prior to randomization and treated with no evidence of disease recurrence and for whom no more than 1 line of chemotherapy was applied.
16. Current active pneumonitis or any history of pneumonitis requiring steroids (any dose) or immunomodulatory treatment within 90 days of planned start of the study.
17. Any clinically significant concomitant disease or condition (such as transfusion-dependent anemia or thrombocytopenia) that could interfere with, or for which the treatment might interfere with, the conduct of the study or that would, in the opinion of the Investigator, pose an unacceptable risk to the patients in this study.
18. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study requirements and/or follow-up procedures. Those conditions should be discussed with the patients before study entry.
19. High medical risk due to a serious, uncontrolled medical disorder; nonmalignant systemic disease; or active, uncontrolled infection (including COVID-19). Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, active uncontrolled coagulopathy, bleeding disorder, or any psychiatric disorder that prohibits obtaining informed consent.
20. Uncontrolled hypertension defined as SBP>180 and DBP>100 should receive antihypertensive medical therapy for blood pressure control (to achieve SBP<160 and DBP <90) before being enrolled in the study.
21. Is pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and/or for up to 180 days after the last dose of study treatment.
22. Presence of hepatitis B surface antigen or a positive hepatitis C virus (HCV) antibody test result at Screening or within 3 months prior to first dose of study treatment. Patients with presence of hepatitis B core antibody should also be excluded.

    1. NOTE: Patients with chronic hepatitis B virus (HBV) infection, who meet the criteria for anti-HBV therapy may be eligible if the participant is on a suppressive antiviral therapy prior to initiation of cancer therapy.
    2. NOTE: Patients with positive HCV antibody due to prior resolved disease can be enrolled only if a confirmatory negative HCV RNA PCR is obtained. Also, patients with a history of HCV infection may be eligible if they have both: completed curative therapy, have an HCV viral load <quantifiable limit.
23. Known history of MDS or AML
24. Are immunocompromised. Patients with splenectomy are allowed. Patients with known human immunodeficiency virus (HIV) are allowed if they meet the following criteria:

    1. Cluster of differentiation 4 ≥350/µL and viral load <400 copies/mL
    2. No history of acquired immunodeficiency syndrome-defining opportunistic infections within 12 months prior to enrollment.
    3. No history of HIV-associated malignancy for the past 5 years. Concurrent antiretroviral therapy as per the most current National Institutes of Health (NIH) Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents Living with HIV [NIH, 2021] started >4 weeks prior to study enrollment.
25. Prior immunotherapy toxicities (until resolution to Grade 1 or better)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 12 months
  Percentage of evaluable patients that experience an objective response (Complete Response (CR) or Partial Response (PR)), per RECISIT v1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Adverse Events Related to Treatment | Up to 12 months
  Rate of Adverse Events (AEs) related to the niraparib and dostarlimab combination per CTCAE v5.0
Progression-free Survival (PFS) | Up to 36 months
  Median time from first response to treatment until documented disease progression by RECIST v1.1 or death due to any cause. Per RECISIT v1.1, Progressive Disease: ≥20%increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Duration of Response (DoR) | Up to 36 months
  Time from first documented response to disease progression by RECIST v1.1 or death in patients who achieve complete or partial response.
Overall Survival (OS) | Up to 36 months
  Time from assignment to treatment arm until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim H Sahin, MD, Principal Investigator — UPMC Hillman Cancer Center

IPD SHARING:
Plan to Share IPD: No